CLINICAL TRIAL: NCT05803486
Title: Correlation Between Quadratus Lumborum , Pelvic Floor Muscles and Diaphragm in Patients With Urinary Incontinence
Status: Completed | Type: Observational
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Other Study IDs: 2\2023
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Correlation Between Quadratus Lumborum , Pelvic Floor Muscles and Diaphragm in Patients With Urinary Incontinence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: examined by ultrasound image to measure quadratus lumborum thickness, pelvic floor muscles force and diaphragm excursion in patients with urinary incontinence
- control group: examined by ultrasound image to measure quadratus lumborum thickness, pelvic floor muscles force and diaphragm excursion in patients with urinary incontinence

SUMMARY:
The purpose of this study is to investigate Correlation between quadratus lumborum , pelvic floor muscles and diaphragm in patients with urinary incontinence

DETAILED DESCRIPTION:
50 patients were distributed randomly into two groups. The first group measured ultrasound imaging for quadratus lumborum , pelvic floor muscles and diaphragm urinary incontinence female The second group measured ultrasound imaging for quadratus lumborum , pelvic floor muscles and diaphragm urinary incontinence female normal females.

Patients examined with medical ultrasound imaging .

ELIGIBILITY:
Inclusion Criteria:

* - Their ages varied from 30to 40years, their body mass index (BMI) was 25-30 kg/m2 and a number of parities ≤ three normal vaginal deliveries, at least two years and Subjects hadn't received drugs , urinary incontinence mild or modrate

Exclusion Criteria:

- 1. History of spinal surgery or spinal fracture. 2. Volunteers with a history of a recto-vaginal or vesico-vaginal fistula, undiagnosed uterine bleeding urinary tract infection, diabetes, intrauterine device, chest and/or cardiac disease and using any drugs for urinary incontinence 3. Serious diseases, such as heart disease, kidney, liver diseases, gastric ulcer or duodenal ulcer.

4. A history of bronchial asthma or any chest disease. 5. Uncontrolled diabetes or hypertension. 6. Patients with peacemaker or any metal implant on the treated area. 7. Cancer or patient with past history of tumor excision.

Ages: 30 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: - Their ages varied from 30to 40years, their body mass index (BMI) was 25-30 kg/m2 and a number of parities ≤ three normal vaginal deliveries, at least two years and Subjects hadn't received drugs
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Force of contraction of pelvic floor muscles | 2 months
  by ultrasound imaging, convex transducer was used at a frequency of 5 MHz for evaluating. Voluntary PFM contractions' force (strength) of all patients.

SECONDARY OUTCOMES:
diaphragm excursion | 2 months
  by ultrasound imaging, convex transducer was used at a frequency of 5 MHz for evaluating. Voluntary diaphragm excursion

OTHER OUTCOMES:
quadratus lumborum thickness | 2 months
  by ultrasound imaging, convex transducer was use quadratus lumborum thickness

CONTACTS AND LOCATIONS:
Overall Officials: doaa A.Nasser abdelhady, Principal Investigator — Deraya University
Locations (1):
- Deraya university, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No